CLINICAL TRIAL: NCT03438110
Title: Project to Understand & Research Preterm Pregnancy Outcomes-South Asia (PURPOSe)
Brief Title: Asia Pregnancy Outcomes Study
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Responsible Party: Principal Investigator, Elizabeth McClure, Senior Research Epidemiologist, RTI International
Other Study IDs: CP COD
Record Dates: First submitted 2018-01-29; First posted 2018-02-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Death; Stillbirth
Keywords: Preterm birth; Neonatal death; Stillbirth; Asia; Africa
MeSH Terms: conditions — Perinatal Death; Stillbirth; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Preterm birth is a major cause of child mortality and morbidity, most of which occurs in south-east Asia and sub-Saharan Africa. To date few neonatal cause of death studies, especially in low- and middle-income countries have determined the specific causes of preterm death, instead attributing all neonatal deaths of infants born at less than 37 weeks to prematurity. Infections are responsible for a large proportion of these deaths but because of complexity and costs associated with testing, little is known about the prevalence of infection-related deaths in preterm infants or the specific pathogens associated with mortality.

The primary objective of this study is to determine the cause of deaths among preterm births and stillbirths. Secondary outcomes include determining the specific pathogens responsible for infection-related deaths, potential preventability of these deaths and interventions which may reduce mortality. One site in India and one in Pakistan will include a total sample size of 700 (350 stillbirths and 350 preterm neonatal deaths) for 1,400 cases to be included in the cause of death analyses. All women who deliver a preterm birth or a stillbirth at the study hospitals will be eligible for inclusion. Among those who consent, an obstetric history, clinical obstetric and (if applicable) neonatal care will be collected as well as research investigations including ultrasound, x-ray, microbiology and minimally invasive tissue sampling and autopsy will be collected.

This study will align with other efforts to determine cause of death among infants and children and ultimately the results will inform future interventions to reduce neonatal mortality and stillbirth. The researchers emphasize that this study, with its focus on preterm neonatal mortality and stillbirth, will provide information not available elsewhere.

DETAILED DESCRIPTION:
Neonatal mortality is common in South Asia and sub-Saharan Africa with rates as high as 40 to 50 per 1,000 live births in some countries compared to rates as low as 2 per 1,000 live births in Scandinavia. Worldwide, at least 2.6 million neonatal deaths occur annually, with more than one-third attributed directly to preterm birth. Globally, the risk of death from preterm birth is highest in south Asia and sub-Saharan Africa. Although the mortality rates are often higher in Africa, numerically, more infants die in south Asia. Preterm neonates die from prematurity-related complications such as respiratory distress syndrome (RDS), necrotizing enterocolitis (NEC), and intraventricular hemorrhage (IVH), and conditions not specifically caused by prematurity such as asphyxia, infection, and congenital anomalies. However, few cause of death studies-especially in low-resource settings in low and middle-income countries (LMIC)-have determined the specific causes of preterm death, instead attributing all neonatal deaths of infants <37 weeks to prematurity. Furthermore, little is known about the causes of death among stillbirths in preterm births in LMIC and especially the specific types of infections associated with stillbirth.

One of the important goals of international organizations is to reduce neonatal mortality in LMIC, with recent efforts highlighting the importance of reducing neonatal mortality in preterm infants. One impeding factor is lack of knowledge about the medical conditions that cause neonatal mortality in preterm infants and the circumstances under which these babies die. It is crucial not only to know the major medical, infectious and pathological causes, but also the sequence of events that led to the death. Answers to these questions are important not only to understand the cause of death in preterm infants, but also to propose effective treatments to reduce the neonatal deaths in live-born preterm infants.

Less is known about the causes of stillbirth than neonatal mortality in LMIC and Asia specifically. Stillbirth rates are also highest in south Asia and sub-Saharan Africa, with rates as high as 40-50/1,000 births compared to 2-3/1,000 in Scandinavia. The highest reported rates of stillbirth occur in Pakistan. In most countries, the stillbirth rates are equivalent to or greater than the neonatal mortality rates with about 3 million third trimester stillbirths occurring yearly. In high-income countries (HIC), 50% of the stillbirths occur prior to 28 weeks and fully 80% occur prior to term. The percent of stillbirths occurring in the preterm period in LMIC is unknown, but probably lower than the HIC rate of 80%, likely in the range of 50%. Thus, the researchers estimate that most the perinatal mortality in LMIC occurs in infants born preterm.

Stillbirths are caused by a variety of maternal and fetal conditions, including placental abruption, obstructed labor, preeclampsia, placental malfunction, infection, congenital anomalies and cord complications, conditions that also contribute to neonatal mortality. The distribution of these causes and the sequence of events leading to the stillbirth in LMIC are generally unknown. One study suggests that when assessing preterm birth, the true picture of preterm birth may be obscured if stillbirth is excluded. In this cross-sectional study of 29 countries, researchers found that inclusion of stillbirths substantially increased the preterm birth rate in all countries. The degree of change was particularly large in LMIC, with the preterm birth rate increasing by 18% when stillbirths were included. Thus, because of the substantial overlap in etiology between preterm neonatal deaths and preterm stillbirths, and the large contribution of stillbirths to the preterm birth rate, the researchers believe that it would be appropriate to evaluate cause of death in all preterm deaths whether live- or stillborn.

For both neonatal deaths and stillbirths, infectious causes of death are often not identified and have largely been under-reported in low-resource settings where both logistics and technology may limit investigations into infections. From a literature review of epidemiological studies and case reports, the list of pathogens potentially causing a stillbirth or neonatal death likely extends to over 100 organisms. Since the identification of pathogens responsible for fetal or neonatal death may not be obtained from blood cultures alone, the identification process becomes more complicated with testing required of specific tissues such as the placenta, and fetal or neonatal organs, often with molecular assays.

In many areas in Asia, most deliveries now occur in health facilities. Despite the dramatic increase in hospital deliveries in the last decade in this region, little reduction in neonatal mortality or stillbirth has been realized. Thus, the Asian study will augment other efforts through examination of the specific causes of preterm neonatal deaths in Asia, and expand understanding of the contribution of preterm birth to perinatal mortality through inclusion of stillbirths. Determining the main causes and risk factors for perinatal mortality will ultimately inform potential strategies to reduce the high neonatal mortality and stillbirth rates currently seen in south Asia. This is a prospective, observational study aimed to better understand causes of stillbirths and neonatal deaths among preterm livebirths in Karachi, Pakistan, and Davengere, India.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor and delivery with imminent preterm delivery and/or stillbirth

Exclusion Criteria:

* Induced (medical) abortion
* Unable to determine the gestational age at delivery
* Gestational age < 20 weeks at delivery

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted at hospitals identified in Karachi, Pakistan and in Davangere, India. All women who deliver a stillbirth and/or who deliver preterm at a study hospital will be screened for study eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 1226 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Cause of Death | At time of study enrollment of mother
  Cause of death among preterm deaths and stillbirths.

SECONDARY OUTCOMES:
Neonatal Death | At time of study enrollment of mother
  Evaluate the rate of mortality by gestational age and birth weight by taking weight post-mortem and estimating gestational age
Preterm Death and Stillbirth Placental Pathology | At time of study enrollment of mother
  Determine the placental pathology associated with stillbirth and preterm deaths by performing post-mortem autopsy
Stillbirth and Preterm Death Pathogens | Following stillbirth or infant death
  Determine the pathogens associated with stillbirth and preterm deaths by examination of samples collected from fetus/neonate at autopsy and maternal samples collected at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McClure, PhD, Principal Investigator — RTI International
Locations (3):
- J.J.M. Medical College Hospitals, Davangere, India
- Pakistan (2):
  - National Institute of Child Health, Karachi, Pakistan
  - Jinnah Postgrad Medical Center, Karachi

REFERENCES:
- [Background] GBD 2015 Child Mortality Collaborators. Global, regional, national, and selected subnational levels of stillbirths, neonatal, infant, and under-5 mortality, 1980-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1725-1774. doi: 10.1016/S0140-6736(16)31575-6. PMID 27733285
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Oza S, Lawn JE, Hogan DR, Mathers C, Cousens SN. Neonatal cause-of-death estimates for the early and late neonatal periods for 194 countries: 2000-2013. Bull World Health Organ. 2015 Jan 1;93(1):19-28. doi: 10.2471/BLT.14.139790. Epub 2014 Nov 17. PMID 25558104
- [Background] Blencowe H, Cousens S, Chou D, Oestergaard M, Say L, Moller AB, Kinney M, Lawn J; Born Too Soon Preterm Birth Action Group. Born too soon: the global epidemiology of 15 million preterm births. Reprod Health. 2013;10 Suppl 1(Suppl 1):S2. doi: 10.1186/1742-4755-10-S1-S2. Epub 2013 Nov 15. PMID 24625129
- [Background] Lackritz EM, Wilson CB, Guttmacher AE, Howse JL, Engmann CM, Rubens CE, Mason EM, Muglia LJ, Gravett MG, Goldenberg RL, Murray JC, Spong CY, Simpson JL; Preterm Birth Research Priority Setting Group. A solution pathway for preterm birth: accelerating a priority research agenda. Lancet Glob Health. 2013 Dec;1(6):e328-30. doi: 10.1016/S2214-109X(13)70120-7. Epub 2013 Nov 15. No abstract available. PMID 25104592
- [Background] McClure EM, Bose CL, Garces A, Esamai F, Goudar SS, Patel A, Chomba E, Pasha O, Tshefu A, Kodkany BS, Saleem S, Carlo WA, Derman RJ, Hibberd PL, Liechty EA, Hambidge KM, Krebs NF, Bauserman M, Koso-Thomas M, Moore J, Wallace DD, Jobe AH, Goldenberg RL. Global network for women's and children's health research: a system for low-resource areas to determine probable causes of stillbirth, neonatal, and maternal death. Matern Health Neonatol Perinatol. 2015 May 4;1:11. doi: 10.1186/s40748-015-0012-7. eCollection 2015. PMID 27057328
- [Background] Engmann C, Jehan I, Ditekemena J, Garces A, Phiri M, Mazariegos M, Chomba E, Pasha O, Tshefu A, Hemed Y, McClure EM, Thorsten V, Bann C, Goldenberg RL, Bose C, Setel P, Carlo WA, Wright LL. Using verbal autopsy to ascertain perinatal cause of death: are trained non-physicians adequate? Trop Med Int Health. 2009 Dec;14(12):1496-504. doi: 10.1111/j.1365-3156.2009.02395.x. Epub 2009 Oct 1. PMID 19799757
- [Background] McClure EM, Garces A, Saleem S, Moore JL, Bose CL, Esamai F, Goudar SS, Chomba E, Mwenechanya M, Pasha O, Tshefu A, Patel A, Dhaded SM, Tenge C, Marete I, Bauserman M, Sunder S, Kodkany BS, Carlo WA, Derman RJ, Hibberd PL, Liechty EA, Hambidge KM, Krebs NF, Koso-Thomas M, Miodovnik M, Wallace DD, Goldenberg RL. Global Network for Women's and Children's Health Research: probable causes of stillbirth in low- and middle-income countries using a prospectively defined classification system. BJOG. 2018 Jan;125(2):131-138. doi: 10.1111/1471-0528.14493. Epub 2017 Jan 31. PMID 28139875
- [Background] Stillbirth Collaborative Research Network Writing Group. Causes of death among stillbirths. JAMA. 2011 Dec 14;306(22):2459-68. doi: 10.1001/jama.2011.1823. PMID 22166605
- [Background] Belizan JM, McClure EM, Goudar SS, Pasha O, Esamai F, Patel A, Chomba E, Garces A, Wright LL, Koso-Thomas M, Moore J, Althabe F, Kodkany BS, Sami N, Manasyan A, Derman RJ, Liechty EA, Hibberd P, Carlo WA, Hambidge KM, Buekens P, Jobe AH, Goldenberg RL. Neonatal death in low- to middle-income countries: a global network study. Am J Perinatol. 2012 Sep;29(8):649-56. doi: 10.1055/s-0032-1314885. Epub 2012 May 29. PMID 22644832
- [Background] Goldenberg RL, McClure EM, Saleem S, Reddy UM. Infection-related stillbirths. Lancet. 2010 Apr 24;375(9724):1482-90. doi: 10.1016/S0140-6736(09)61712-8. Epub 2010 Mar 9. PMID 20223514
- [Background] Castillo P, Ussene E, Ismail MR, Jordao D, Lovane L, Carrilho C, Lorenzoni C, Lacerda MV, Palhares A, Rodriguez-Carunchio L, Martinez MJ, Vila J, Bassat Q, Menendez C, Ordi J. Pathological Methods Applied to the Investigation of Causes of Death in Developing Countries: Minimally Invasive Autopsy Approach. PLoS One. 2015 Jun 30;10(6):e0132057. doi: 10.1371/journal.pone.0132057. eCollection 2015. PMID 26126191
- [Background] Jehan I, Harris H, Salat S, Zeb A, Mobeen N, Pasha O, McClure EM, Moore J, Wright LL, Goldenberg RL. Neonatal mortality, risk factors and causes: a prospective population-based cohort study in urban Pakistan. Bull World Health Organ. 2009 Feb;87(2):130-8. doi: 10.2471/blt.08.050963. PMID 19274365
- [Background] McClure EM, Goldenberg RL, Jobe AH, Miodovnik M, Koso-Thomas M, Buekens P, Belizan J, Althabe F. Reducing neonatal mortality associated with preterm birth: gaps in knowledge of the impact of antenatal corticosteroids on preterm birth outcomes in low-middle income countries. Reprod Health. 2016 May 24;13(1):61. doi: 10.1186/s12978-016-0180-6. PMID 27221397
- [Background] Saleem S, Reza T, McClure EM, Pasha O, Moss N, Rouse DJ, Bartz J, Goldenberg RL. Chlorhexidine vaginal and neonatal wipes in home births in Pakistan: a randomized controlled trial. Obstet Gynecol. 2007 Nov;110(5):977-85. doi: 10.1097/01.AOG.0000285653.17869.26. PMID 17978107
- [Background] Saleem S, Rouse DJ, McClure EM, Zaidi A, Reza T, Yahya Y, Memon IA, Khan NH, Memon G, Soomro N, Pasha O, Wright LL, Moore J, Goldenberg RL. Chlorhexidine vaginal and infant wipes to reduce perinatal mortality and morbidity: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1225-1232. doi: 10.1097/AOG.0b013e3181e00ff0. PMID 20502294
- [Background] Goudar SS, Goco N, Somannavar MS, Vernekar SS, Mallapur AA, Moore JL, Wallace DD, Sloan NL, Patel A, Hibberd PL, Koso-Thomas M, McClure EM, Goldenberg RL. Institutional deliveries and perinatal and neonatal mortality in Southern and Central India. Reprod Health. 2015;12 Suppl 2(Suppl 2):S13. doi: 10.1186/1742-4755-12-S2-S13. Epub 2015 Jun 8. PMID 26063586
- [Background] Pasha O, Saleem S, Ali S, Goudar SS, Garces A, Esamai F, Patel A, Chomba E, Althabe F, Moore JL, Harrison M, Berrueta MB, Hambidge K, Krebs NF, Hibberd PL, Carlo WA, Kodkany B, Derman RJ, Liechty EA, Koso-Thomas M, McClure EM, Goldenberg RL. Maternal and newborn outcomes in Pakistan compared to other low and middle income countries in the Global Network's Maternal Newborn Health Registry: an active, community-based, pregnancy surveillance mechanism. Reprod Health. 2015;12 Suppl 2(Suppl 2):S15. doi: 10.1186/1742-4755-12-S2-S15. Epub 2015 Jun 8. PMID 26062610
- [Background] Goldenberg RL, Gravett MG, Iams J, Papageorghiou AT, Waller SA, Kramer M, Culhane J, Barros F, Conde-Agudelo A, Bhutta ZA, Knight HE, Villar J. The preterm birth syndrome: issues to consider in creating a classification system. Am J Obstet Gynecol. 2012 Feb;206(2):113-8. doi: 10.1016/j.ajog.2011.10.865. Epub 2011 Oct 25. PMID 22177186
- [Background] Goldenberg RL, McClure EM, Jobe AH, Kamath-Rayne BD, Gravette MG, Rubens CE. Stillbirths and neonatal mortality as outcomes. Int J Gynaecol Obstet. 2013 Dec;123(3):252-3. doi: 10.1016/j.ijgo.2013.06.020. Epub 2013 Sep 4. PMID 24050480
- [Background] Dudley DJ, Goldenberg R, Conway D, Silver RM, Saade GR, Varner MW, Pinar H, Coustan D, Bukowski R, Stoll B, Koch MA, Parker CB, Reddy UM; Stillbirth Research Collaborative Network. A new system for determining the causes of stillbirth. Obstet Gynecol. 2010 Aug;116(2 Pt 1):254-260. doi: 10.1097/AOG.0b013e3181e7d975. PMID 20664383
- [Background] Garces AL, McClure EM, Perez W, Hambidge KM, Krebs NF, Figueroa L, Bose CL, Carlo WA, Tenge C, Esamai F, Goudar SS, Saleem S, Patel AB, Chiwila M, Chomba E, Tshefu A, Derman RJ, Hibberd PL, Bucher S, Liechty EA, Bauserman M, Moore JL, Koso-Thomas M, Miodovnik M, Goldenberg RL. The Global Network Neonatal Cause of Death algorithm for low-resource settings. Acta Paediatr. 2017 Jun;106(6):904-911. doi: 10.1111/apa.13805. Epub 2017 Apr 5. PMID 28240381
- [Derived] McClure EM, Saleem S, Goudar SS, Dhaded S, Guruprasad G, Kumar Y, Tikmani SS, Kadir M, Raza J, Yasmin H, Moore JL, Kim J, Bann C, Parlberg L, Aceituno A, Carlo WA, Silver RM, Lamberti L, Patterson J, Goldenberg RL. The project to understand and research preterm pregnancy outcomes and stillbirths in South Asia (PURPOSe): a protocol of a prospective, cohort study of causes of mortality among preterm births and stillbirths. Reprod Health. 2018 Jun 22;15(Suppl 1):89. doi: 10.1186/s12978-018-0528-1. PMID 29945651